CLINICAL TRIAL: NCT03076450
Title: Clinical Evaluation of Point-of-care Lung Ultrasound Combined With Pressure-volume Curve to Titration Adjust PEEP for ARDS Lung Recruitment
Brief Title: Evaluation of POC Lung Ultrasound Combined With Pressure-volume Curve to Titration Adjust PEEP for ARDS Lung Recruitment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pudong New Area Gongli Hospital (Other)
Collaborators: Shanghai Municipal Commission of Health and Family Planning (Other)
Responsible Party: Principal Investigator, Qiancheng Luo, Attending-doctor of Critical Care Medcine, Principal Investigator, Shanghai Pudong New Area Gongli Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201640405
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome, ARDS; Point-of-care lung ultrasound,POC-LUS; Pressure-volume curve, PVC; Positive end-expiratory pressure, PEEP; Ultrasound re-aeration score, US-RAS
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventricular Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maximum Oxygenation (Active Comparator): Using PVC to set the initial peep, check ABG real-time, and according to PaO2+PaCO2≥400mmHg whether or not to adjust maintain PEEP.
  Interventions: Diagnostic Test: Maximum Oxygenation
- Lung Ultrasound Re-aeration Score (Experimental): Combine POC-LUS with PVC in set the initial peep, and then dynamic record LUS-RAS to feedback regulate PEEP.
  Interventions: Device: Lung Ultrasound

INTERVENTIONS:
Device: Lung Ultrasound — Adjust PEEP real-time in term of LUS-RAS chang.
  Arms: Lung Ultrasound Re-aeration Score
Diagnostic Test: Maximum Oxygenation — Adjust PEEP real-time in term of PaO2+PaCO2≥400mmHg whether or not.
  Arms: Maximum Oxygenation

SUMMARY:
Using lung ultrasound re-aeration score(LUS-RAS) combined with pressure-volume curve(PVC) adjust maintain positive end-expiratory pressure(PEEP) after recruitment maneuver, to achieve real-time adjustment, reduce ventilation-associated lung injury and the purpose of effective lung recruitment.

DETAILED DESCRIPTION:
The traditional method, set PEEP according to PVC in ARDS mechanical ventilation, lacks morphological evaluation. For point-of-care lung ultrasound(POC-LUS) is non-invasive, real-time, visualization, no need transport patients, getting more and more attention in the ARDS treatment. It has been reported that LUS-RAS is a meaningful assessment in recruitment maneuver. This study will combine POC-LUS with PVC in set the initial peep, and then dynamic record LUS-RAS to feedback regulate PEEP. Using the POC-LUS and maximum oxygenation method to assess lung recruitment effect in experimental group and control group prospectively. The ventilator parameters, state of hemodynamic, arterial blood gas(ABG) in each group will be recorded; Statistical methods will be performed in term to understand the correlation.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18 years and older
* ARDS patients with invasive mechanical ventilation

Exclusion Criteria:

* Intracranial hypertension
* Pneumothorax and mediastinal emphysema
* Severe hypoxemia (oxygenation index <100)
* Hemodynamic instability
* Chest deformity or surgical history
* Affect Lung-ultrasound conditions: subcutaneous emphysema, chest wound etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Lung Ultrasound re-aeration score, LUS-RAS | 48 hours
  The score is composed of 12 different regions of chest wall checked by POC-LUS.

CONTACTS AND LOCATIONS:
Overall Officials: Qiancheng Luo, MM, Principal Investigator — Shanghai Pudong New Area Gongli Hospital
Locations (1):
- Gongli Hospital, Pudong, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes